CLINICAL TRIAL: NCT04458194
Title: A Feasibility Trial Comparing the Effectiveness of Virtual YOCAS©® Yoga to Standard Care for Treating Insomnia in Cancer Survivors
Brief Title: Comparing Virtual Yoga to Standard Care on Insomnia Among Cancer Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Bassett Medical Center (Other)
Responsible Party: Principal Investigator, Karen Mustian, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY00004405
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Care (Active Comparator): Cancer survivors receive their standard care
  Interventions: Other: Standard Care
- YOCAS (Experimental): Cancer survivors receive 8 virtual yoga sessions (75 minutes/session, 2 times a week for 4 weeks) delivered via an electronic platform (e.g., Zoom)
  Interventions: Behavioral: YOCAS©® yoga

INTERVENTIONS:
Other: Standard Care — Standard Care is used as a control condition. Cancer survivors assigned to this arm continue to receive standard care from their medical providers.
  Arms: Standard Care
Behavioral: YOCAS©® yoga — Yoga for Cancer Survivors, YOCAS©®, intervention is a low to moderate intensity mode of exercise that draws from two basic types of yoga; gentle Hatha and Restorative yoga. The program includes specific physical postures and mindfulness exercises focused on breathing and meditation. Cancer survivors will participate in 8 virtual YOCAS sessions (75 minutes/session, 2 times a week for 4 weeks) delivered via an electronic platform (e.g., Zoom)
  Arms: YOCAS

SUMMARY:
This feasibility phase II randomized controlled trial examines the preliminary efficacy of our standardized four-week YOCAS©® (Yoga for Cancer Survivors) intervention that is delivered virtually on insomnia and sleep quality in cancer survivors.

Insomnia can be described as excessive daytime napping, difficulty falling asleep, difficulty staying asleep, or waking up earlier than desired. The vast majority of patients with cancer experience some form of sleep impairment post-treatment. Yoga is safe, feasible, and effective for improving insomnia and sleep quality in cancer survivors. However, most of the yoga intervention was delivered in person. With the challenges and the social distancing regulation regarding the COVID-19 pandemic, adapting to virtual behavioral intervention is critically important and needed. Whether the yoga intervention delivered virtually to survivors provides a similar benefit of improving insomnia and sleep quality is unknown.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To compare the effects of virtual YOCAS©® intervention to standard care on changes in insomnia measured via the Insomnia Severity Index among cancer survivors

SECONDARY OBJECTIVE:

To compare the effects of virtual YOCAS©® intervention to standard care on changes in sleep quality measured via the Pittsburgh Sleep Quality Index among cancer survivors

OUTLINE: Cancer survivors are randomized to 1 of 2 arms.

ARM I: Standard Care: Cancer survivors receive their standard care

ARM II: YOCAS©® intervention: Cancer survivors participate in 8 virtual YOCAS sessions (75 minutes/session, 2 times a week for 4 weeks) delivered via the electronic platform (e.g., Zoom)

ELIGIBILITY:
Inclusion Criteria:

Cancer Survivors must:

* have a confirmed diagnosis of cancer
* have received surgery, chemotherapy, and/or radiation therapy
* have completed all surgery, chemotherapy, and/or radiation therapy within the last 2 months to 10 years
* score ≥4 on a 0-10 sleep screening scale
* be at least 18 years of age
* be able to read and understand English
* be able to provide informed consent
* have access to the internet and a smartphone, tablet, and/or computer
* have the ability to attend 8 virtual yoga sessions

Exclusion Criteria:

Cancer Survivor must not:

* have contraindications to yoga participation
* have practiced yoga within the 3 months prior to enrolling in the study
* be planning to start yoga on their own during the time they are enrolled in the study
* have a confirmed diagnosis of sleep apnea or restless leg syndrome
* be receiving any form of treatment for cancer with the exception of hormonal or biologic therapy
* have distant metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-01-12 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Mean change in insomnia as measured by the Insomnia Severity Index (ISI) total score comparing cancer survivors in YOCAS vs. Standard Care | baseline to week 5
  The Insomnia Severity Index is a validated measure of insomnia. A 5-point Likert scale of 7 questions is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28 with higher scores indicating higher severity of insomnia. A linear mixed effects ANCOVA will be used to assess the statistical significance of the differences in mean change among cancer survivors in YOCAS vs. Standard Care

SECONDARY OUTCOMES:
Mean Change in sleep quality as measured by the Pittsburgh Sleep Quality Inventory (PSQI) total Score comparing cancer survivors in YOCAS vs. Standard Care | baseline to week 5
  The PSQI measures sleep quality with a total score ranging from 0-21 with higher scores indicating worse sleep quality. A linear mixed effects ANCOVA will be used to assess the statistical significance of the differences in mean change among cancer survivors in YOCAS vs. Standard Care

CONTACTS AND LOCATIONS:
Overall Officials: Karen Mustian, PhD, MPH, Principal Investigator — University of Rochester
Locations (2):
- United States (2):
  - Bassett Research Institute, Cooperstown, New York
  - University of Rochester Medical Center, Rochester, New York

IPD SHARING:
Plan to Share IPD: No